CLINICAL TRIAL: NCT07305103
Title: Defining Dosimetric Reference Levels in Computed Tomography Spectral Scanning
Acronym: NR Spectral
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut Paoli Calmettes, Marseille (Unknown); Hôpital Necker-Enfants Malades (Other); Lille University Hospital (Unknown); CHU Hôpital Lariboisière APHP (Unknown); Centre Hospitalier Universitaire de Saint Etienne (Other); Saint-Louis Hospital, Paris, France (Other); Bichat Hospital (Other); Hôpital Louis Mourier, 92700 Colombes (Unknown); Centre Hospitalier de Valenciennes (Network); Hopital Louis Pradel (Other); Centre Léon Bérard, Lyon (Unknown); University Hospital, Bordeaux (Other); Centre Hospitalier Lyon Sud (Other); Institut Curie (Other); Amiens University Hospital (Other); Poitiers University Hospital (Other); Henri Mondor Hospital, Créteil (Unknown); Saint Antoine University Hospital (Other); Nord Ardennes Intercommunal Hospital (Unknown); Centre Antoine Lacassagne, Nice (Unknown); Hôpital Edouard Herriot (GH Centre), Lyon (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2024-1/DD-01
Record Dates: First submitted 2025-09-10; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Medical Imaging
Keywords: Radiation dose; Reference levels; Radiology; Spectral Computed Tomography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing a maximum number of 18 spectral CT scans among the examinations mentioned below: Patients undergoing a maximum number of 18 spectral CT scans among the examinations mentioned below:
  1. Chest CT for pulmonary embolism
  2. Chest CT for other indications
  3. Coronary CT with contrast injection and retrospective gating
  4. Coronary CT with contrast injection and prospective gating
  5. Cranial CT with contrast injection
  6. Supra-aortic trunk CT
  7. Neck and ear,nose and throat sphere CT with contrast injection
  8. Oncological abdomen-pelvis CT scan
  9. Abdomen-pelvis CT scan to check for kidney stones
  10. Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones
  11. Oncological chest-abdomen-pelvis CT scan
  12. Non-oncological chest-abdomen-pelvis CT scan
  13. Oncological chest-abdomen CT scan
  14. Non-oncological chest-abdomen CT scan
  15. Lower limb angiography
  16. Cervical spine CT scan
  17. Thoracic spine CT scan
  18. Lumbar spine CT scan
  19. Pelvis CT scan,
  20. Extremities CT scan
  Interventions: Radiation: Spectral ComputedTomography

INTERVENTIONS:
Radiation: Spectral ComputedTomography — Commonly performed spectral computed tomography examinations in France

SUMMARY:
Spectral computed tomography or dual-energy CT imaging can overcome the limitations of conventional CT in differentiating between two materials with equivalent total attenuation. It can generate several types of images, such as virtual monochromatic images, which improve the contrast-to-noise ratio for low energy levels and reduce artifacts for high energy levels. It also allows for quantitative image analysis and thus better characterization of lesions and tissues through material mapping (e.g., iodinated contrast agent mapping). This technique is increasingly used in routine clinical practice thanks to improvements in image flow management and technological advances. It also involves exposing patients to ionizing radiation, as with conventional CT but, unlike conventional CT scans, for which dosimetric reference levels (RLs) are defined for the most common examinations in France (RL decree dated 2019), there are currently no dosimetric reference levels for examinations performed using this technique. Yet RLs are an important and effective tools for optimizing patient exposure to ionizing radiation. Several articles were published between 2012 and 2017 when the first dual-energy scanners arrived in clinics. However, the results presented in these studies are now far removed from recent practices, as they do not take into account the latest technological developments used in dual-energy scanners, which reduce X-ray doses.

The main objective of the study is to define dosimetric reference levels for the most commonly performed spectral computed tomography examinations in France.

DETAILED DESCRIPTION:
Spectral computed tomography (CT) (or dual-energy CT) imaging can overcome the limitations of conventional CT in differentiating between two materials with equivalent total attenuation. It can generate several types of images, such as virtual monochromatic images, which improve the contrast-to-noise ratio for low energy levels and reduce artifacts for high energy levels. It also allows for quantitative image analysis and thus better characterization of lesions and tissues through material mapping (e.g., iodinated contrast agent mapping). This technique is increasingly used in routine clinical practice thanks to improvements in image flow management and technological advances. It also involves exposing patients to ionizing radiation, as with conventional CT.

However, unlike conventional CT scans, for which dosimetric reference levels (RLs) are defined for the most common examinations in France (RL decree dated 2019), there are currently no dosimetric reference levels for examinations performed using this technique. Yet the RL is an important and effective tool in optimizing patient exposure to ionizing radiation. In fact, a number of articles were published between 2012 and 2017, when the first dual-energy scanners arrived in clinics. However, the results presented in these studies are now far removed from recent practices, as they do not take into account the latest technological developments used in dual-energy scanners, which reduce X-ray doses.

The main objective of the study is to define dosimetric reference levels for the most frequently performed spectral computed tomography examinations in France:

1. Chest CT for pulmonary embolism
2. Chest CT for other indications
3. Coronary CT with contrast injection and retrospective gating
4. Coronary CT with contrast injection and prospective gating
5. Cranial CT with contrast injection
6. Supra-aortic trunk CT
7. Neck and ear,nose and throat sphere CT with contrast injection
8. Oncological abdomen-pelvis CT scan
9. Abdomen-pelvis CT scan to check for kidney stones
10. Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones
11. Oncological chest-abdomen-pelvis CT scan
12. Non-oncological chest-abdomen-pelvis CT scan
13. Oncological chest-abdomen CT scan
14. Non-oncological chest-abdomen CT scan
15. Lower limb angiography
16. Cervical spine CT scan
17. Thoracic spine CT scan
18. Lumbar spine CT scan
19. Pelvis CT scan,
20. Extremities CT scan

The secondary objectives of the study are to evaluate, for each examination performed:

1. the impact of the spectral acquisition/detection technique on the dose delivered to patients.
2. the impact of patients' BMI on the dose delivered to patients.
3. the impact of reconstruction algorithms on the dose delivered to patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male/female patient (≥ 18 years old)
* Body Mass Index (BMI) between 18 and 35 kg/m²
* Patients who underwent a spectral CT scan between January 1, 2023, and August 31, 2024, as part of their treatment.

Exclusion Criteria:

- Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent a spectral CT scan between January 1, 2023, and August 31, 2024, as part of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 9600 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dosimetric reference levels for spectral computed tomography examinations in France: Chest CT for pulmonary embolism. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Chest CT for pulmonary embolism. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Chest CT for other indications. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Chest CT for other indications. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Coronary CT with contrast injection and retrospective gating. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Coronary CT with contrast injection and prospective gating. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Cranial CT with contrast injection. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Cranial CT with contrast injection. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Supra-aortic trunk CT. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Supra-aortic trunk CT. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Neck and ear,nose and throat sphere CT with contrast injection. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Neck and ear,nose and throat sphere CT with contrast injection. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological abdomen-pelvis CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological abdomen-pelvis CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Abdomen-pelvis CT scan to check for kidney stones. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Abdomen-pelvis CT scan to check for kidney stones. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological chest-abdomen-pelvis CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological chest-abdomen-pelvis CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Non-oncological chest-abdomen-pelvis CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Non-oncological chest-abdomen-pelvis CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological chest-abdomen CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Oncological chest-abdomen CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Non-oncological chest-abdomen CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Non-oncological chest-abdomen CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Lower limb angiography. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Lower limb angiography. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Cervical spine CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Cervical spine CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Thoracic spine CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Thoracic spine CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Lumbar spine CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Lumbar spine CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Pelvis CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Pelvis CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm
Dosimetric reference levels for spectral computed tomography examinations in France: Extremities CT scan. CTDIvol | Periprocedural
  Computed tomography dose index (CTDIvol) per acquisition expressed in milligray (mGy).
Dosimetric reference levels for spectral computed tomography examinations in France: Extremities CT scan. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm will be recorded

SECONDARY OUTCOMES:
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for pulmonary embolism. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for pulmonary embolism. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for pulmonary embolism. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for pulmonary embolism. DLP | Periprocedural
  Dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients: Chest CT for pulmonary embolism. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients: Chest CT for pulmonary embolism. Acquisition parameters, kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients: Chest CT for pulmonary embolism. Acquisition parameters, mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients: Chest CT for pulmonary embolism. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients: Chest CT for pulmonary embolism. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Chest CT for pulmonary embolism. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for other indications. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for other indications. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for other indications. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Chest CT for other indications. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients: Chest CT for other indications. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients: Chest CT for other indications. Acquisition parameters, kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients: Chest CT for other indications. Acquisition parameters, mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients: Chest CT for other indications. Acquisition parameters, rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients: Chest CT for other indications. Acquisition parameters, helical pitch | Periprocedural
  Helical pitch time will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Chest CT for other indications. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Coronary CT with contrast injection and retrospective gating. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Coronary CT with contrast injection and retrospective gating. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Coronary CT with contrast injection and retrospective gating. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Coronary CT with contrast injection and retrospective gating. DLP | Periprocedural
  The dose length product (DLP) will be recorded.
Impact of patients' BMI on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. Acquisition parameters, kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. Acquisition parameters, mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Coronary CT with contrast injection and retrospective gating. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cranial CT with contrast injection. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cranial CT with contrast injection. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cranial CT with contrast injection. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cranial CT with contrast injection. DLP | Periprocedural
  Dose length product (DLP) will be recorded.
Impact of patients' BMI on the dose delivered to patients: Cranial CT with contrast injection. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients: Cranial CT with contrast injection. Acquisition parameters, kV | Periprocedural
  Acquisition parameters (kV)will be recorded
Impact of patients' BMI on the dose delivered to patients: Cranial CT with contrast injection. Acquisition parameters, mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients: Cranial CT with contrast injection. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients: Cranial CT with contrast injection. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Cranial CT with contrast injection. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Supra-aortic trunk CT. Acquisition type | Periprocedural
  The type of acquisition will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Supra-aortic trunk CT. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Supra-aortic trunk CT. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Supra-aortic trunk CT. DLP | Periprocedural
  The dose (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Supra-aortic trunk CT. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Supra-aortic trunk CT. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Supra-aortic trunk CT. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Supra-aortic trunk CT. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Supra-aortic trunk CT. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Neck and ear, nose and throat sphere CT with contrast injection. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Neck and ear, nose and throat sphere CT with contrast injection. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Neck and ear, nose and throat sphere CT with contrast injection. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Neck and ear, nose and throat sphere CT with contrast injection. DLP | Periprocedural
  The dose (DLP) expressed in mGy.cm will be recorded
Impact of patients' BMI on the dose delivered to patients : Neck and ear, nose and throat sphere CT with contrast injection. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of reconstruction algorithms on the dose delivered to patients : Neck and ear, nose and throat sphere CT with contrast injection. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological abdomen-pelvis CT scan. Acquisition type | Periprocedural
  The type of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological abdomen-pelvis CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological abdomen-pelvis CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological abdomen-pelvis CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological abdomen-pelvis CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Oncological abdomen-pelvis CT scan. Acquisition parameters (kV) | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological abdomen-pelvis CT scan. Acquisition parameters (mAs) | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological abdomen-pelvis CT scan. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Oncological abdomen-pelvis CT scan. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients: Oncological abdomen-pelvis CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan to check for kidney stones. Acquisition type an | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan to check for kidney stones. Number of acquisitions an | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan to check for kidney stones. CTDIvol an | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan to check for kidney stones. DLP an | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. BMI an | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. Acquisition parameters. Kv an | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. Acquisition parameters. mAs an | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. Rotation time an | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. Helical pitch an | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Abdomen-pelvis CT scan to check for kidney stones. Type of reconstruction algorithm an | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Abdomen-pelvis CT scan for non-oncological purposes and to check for kidney stones. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen-pelvis CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen-pelvis CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen-pelvis CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen-pelvis CT scan. DLP | Periprocedural
  The dose (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Oncological chest-abdomen-pelvis CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen-pelvis CT scan. Acquisition type. | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen-pelvis CT scan. Number of acquisitions. | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen-pelvis CT scan. CDTIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen-pelvis CT scan. CDTIvol. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Non-oncological chest-abdomen-pelvis CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen CT scan. Aquisition type | Periprocedural
  The type of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen CT scan. Number of aquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen CT scan. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Oncological chest-abdomen CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen CT scan. Acquisition parameters (kV) | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen CT scan. Acquisition parameters (mAs) | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen CT scan. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Oncological chest-abdomen CT scan. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Oncological chest-abdomen CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Non-oncological chest-abdomen CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen CT scan | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Non-oncological chest-abdomen CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of reconstruction algorithms on the dose delivered to patients: Non-oncological chest-abdomen CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. Number of acquitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. CTDIvol | Periprocedural
  The dose CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Lower limb angiography. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Lower limb angiography. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Lower limb angiography. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. Rotation time | Periprocedural
  Rotation time will be recorded in seconds.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio.This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lower limb angiography. Type of reconstruction algorithm | Periprocedural
  Type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cervical spine CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cervical spine CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cervical spine CT scan. CDTIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Cervical spine CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Cervical spine CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Cervical spine CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Cervical spine CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Cervical spine CT scan. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Cervical spine CT scan. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Cervical spine CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Thoracic spine CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Thoracic spine CT scan. Number of acquisitions | Periprocedural
  The number of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Thoracic spine CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Thoracic spine CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Thoracic spine CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Thoracic spine CT scan. Acquisition parameters (kV) | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Thoracic spine CT scan. Acquisition parameters (mAs) | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Thoracic spine CT scan. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Thoracic spine CT scan. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Thoracic spine CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lumbar spine CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lumbar spine CT scan. Number of acquisitions | Periprocedural
  The number of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lumbar spine CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Lumbar spine CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded
Impact of patients' BMI on the dose delivered to patients : Lumbar spine CT scan. BMI | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Lumbar spine CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Lumbar spine CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Lumbar spine CT scan. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Lumbar spine CT scan. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients: Lumbar spine CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Pelvis CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Pelvis CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Pelvis CT scan. CTDIvol | Periprocedural
  The dose (CDTIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Pelvis CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded.
Impact of patients' BMI on the dose delivered to patients : Pelvis CT scan. BMI. | Periprocedural
  Weight and height will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Pelvis CT scan. Acquistion parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Pelvis CT scan. Acquistion parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Pelvis CT scan. Acquistion parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Pelvis CT scan. Acquistion parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients : Pelvis CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Extremities CT scan. Acquisition type | Periprocedural
  The type of acquisition will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Extremities CT scan. Number of acquisitions | Periprocedural
  The number of acquisitions will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Extremities CT scan. CTDIvol | Periprocedural
  The dose (CTDIvol) will be recorded.
Impact of the spectral acquisition/detection technique on the dose delivered to patients: Extremities CT scan. DLP | Periprocedural
  The dose length product (DLP) expressed in mGy.cm will be recorded
Impact of patients' BMI on the dose delivered to patients : Extremities CT scan. BMI | Periprocedural
  Weight in kg and height in cm in will be combined to report BMI in kg/m^2
Impact of patients' BMI on the dose delivered to patients : Extremities CT scan. Acquisition parameters. kV | Periprocedural
  Acquisition parameters (kV) will be recorded
Impact of patients' BMI on the dose delivered to patients : Extremities CT scan. Acquisition parameters. mAs | Periprocedural
  Acquisition parameters (mAs) will be recorded
Impact of patients' BMI on the dose delivered to patients : Extremities CT scan. Acquisition parameters. Rotation time | Periprocedural
  Rotation time will be recorded in seconds
Impact of patients' BMI on the dose delivered to patients : Extremities CT scan. Acquisition parameters. Helical pitch | Periprocedural
  Helical pitch will be recorded as a ratio. This represents the relationship between patient couch movement and X-ray beam width. It is the distance travelled by the table during one 360 degree gantry rotation divided by the collimated section thickness
Impact of reconstruction algorithms on the dose delivered to patients: Extremities CT scan. Type of reconstruction algorithm | Periprocedural
  The type of reconstruction algorithm (iterative or deep learning) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Joël GREFFIER, Study Chair — Nîmes University Hospital
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Henzler T, Fink C, Schoenberg SO, Schoepf UJ. Dual-energy CT: radiation dose aspects. AJR Am J Roentgenol. 2012 Nov;199(5 Suppl):S16-25. doi: 10.2214/AJR.12.9210. PMID 23097163
- [Background] Ghasemi Shayan R, Oladghaffari M, Sajjadian F, Fazel Ghaziyani M. Image Quality and Dose Comparison of Single-Energy CT (SECT) and Dual-Energy CT (DECT). Radiol Res Pract. 2020 Apr 20;2020:1403957. doi: 10.1155/2020/1403957. eCollection 2020. PMID 32373363
- [Background] Greffier J, Villani N, Defez D, Dabli D, Si-Mohamed S. Spectral CT imaging: Technical principles of dual-energy CT and multi-energy photon-counting CT. Diagn Interv Imaging. 2023 Apr;104(4):167-177. doi: 10.1016/j.diii.2022.11.003. Epub 2022 Nov 19. PMID 36414506
- [Background] Dabli D, Frandon J, Belaouni A, Akessoul P, Addala T, Berny L, Beregi JP, Greffier J. Optimization of image quality and accuracy of low iodine concentration quantification as function of dose level and reconstruction algorithm for abdominal imaging using dual-source CT: A phantom study. Diagn Interv Imaging. 2022 Jan;103(1):31-40. doi: 10.1016/j.diii.2021.08.004. Epub 2021 Oct 6. PMID 34625394
- [Background] Si-Mohamed SA, Boccalini S, Villien M, Yagil Y, Erhard K, Boussel L, Douek PC. First Experience With a Whole-Body Spectral Photon-Counting CT Clinical Prototype. Invest Radiol. 2023 Jul 1;58(7):459-471. doi: 10.1097/RLI.0000000000000965. Epub 2023 Feb 22. PMID 36822663
- [Background] Wortman JR, Shyu JY, Dileo J, Uyeda JW, Sodickson AD. Dual-energy CT for routine imaging of the abdomen and pelvis: radiation dose and image quality. Emerg Radiol. 2020 Feb;27(1):45-50. doi: 10.1007/s10140-019-01733-9. Epub 2019 Nov 1. PMID 31673838
- [Background] Noda Y, Kawai N, Kawamura T, Kobori A, Miyase R, Iwashima K, Kaga T, Miyoshi T, Hyodo F, Kato H, Matsuo M. Radiation and iodine dose reduced thoraco-abdomino-pelvic dual-energy CT at 40 keV reconstructed with deep learning image reconstruction. Br J Radiol. 2022 Jun 1;95(1134):20211163. doi: 10.1259/bjr.20211163. Epub 2022 Mar 4. PMID 35230135
- [Background] Etard C, Bigand E, Salvat C, Vidal V, Beregi JP, Hornbeck A, Greffier J. Patient dose in interventional radiology: a multicentre study of the most frequent procedures in France. Eur Radiol. 2017 Oct;27(10):4281-4290. doi: 10.1007/s00330-017-4780-5. Epub 2017 Mar 13. PMID 28289939
- [Background] Greffier J, Ferretti G, Rousseau J, Andreani O, Alonso E, Rauch A, Gillet R, Le Roy J, Cabrol-Faivre L, Douane F, David A, Henry S, Jacques T, Stefanovic X, Decoux E, Lafay F, Pilleul F, Couzon F, Boutet C, Woerly B, Baur P, Sans N, Faruch M, Moussier-Lherm A, Tselikas L, Jacquier A, Bigand E, Pessis E, Teriitehau C, Magnier F, Cassagnes L, Haberlay M, Boutteau D, De Kerviler E, Majorel-Gouthain C, Defez D, Vuillod A, Rouviere O, Hennequin L, Fohlen A, Alwan R, Malakhia A, Aubry S, Dohan A, Eresue-Bony M, Gautier R, Dal R, Dabli D, Hebert T, Kovacs R, Hadid-Beurrier L, Bousson V, Potel M, Barbotteau Y, Michel C, Habib-Geryes B, Andre M, Arnaud T, Bestion N, Ernst O, Monfraix S, Brillet PY, Guiu B, Boussel L, Demonchy M, Beregi JP, Frandon J. National dose reference levels in computed tomography-guided interventional procedures-a proposal. Eur Radiol. 2020 Oct;30(10):5690-5701. doi: 10.1007/s00330-020-06903-9. Epub 2020 May 2. PMID 32361774